CLINICAL TRIAL: NCT04911972
Title: Functional Muscle Transfers to Restore Normal Function After Major Lower Limb Sarcoma/ Trauma - Assessment by Gait Analysis and Virtual Reality Environmental Simulation
Brief Title: Functional Muscle Transfers in Lower Limb Sarcoma: 3D Gait Analysis and Environmental Simulation
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Strathclyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN17OR618
Record Dates: First submitted 2021-05-15; First posted 2021-06-03 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Sarcoma; Muscle Tumor; Muscle Loss
MeSH Terms: conditions — Sarcoma; Muscle Neoplasms; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Functional muscle transfer group: Patients who have undergone functional muscle transfer to restore function after tumour surgery or injury, in which the tumour surgery or injury has resulted in functional loss.
  Interventions: Procedure: Functional muscle transfer
- Non-functional muscle transfer group: Patients who have not undergone functional muscle transfer to restore function after tumour surgery or injury, in which the tumour surgery or injury has resulted in functional loss.

INTERVENTIONS:
Procedure: Functional muscle transfer — Muscle transfer to restore lower limb function
  Groups: Functional muscle transfer group

SUMMARY:
The purpose of this study is to assess patient's function after functional limb restoring surgery, performed after ablative tumour surgery or trauma. However, there are no studies as yet providing objective proof of the recovery of function after this type of surgery. This study will use 3D Gait Analysis, Environmental simulation and Patient Reported Outcome Measures to compare patients with function restoring surgery against patients without function restoring surgery.

DETAILED DESCRIPTION:
Introduction

Rationale

The purpose of this study is to assess patient's function after functional limb restoring surgery, performed after ablative tumour surgery or trauma. However, there are no studies as yet providing objective proof of the recovery of function after this type of surgery.

Background information including literature review

Sarcoma surgery has progressed from limb amputation to limb preserving surgery since the early 1980s. Although this has been a major advance, a preserved limb does not equate to a functional limb. Patients may be left with significant disability and reliant on walking aids or braces, and unable to return to normal activities

The West of Scotland Sarcoma service has developed and refined surgical procedures to restore function in the lower limb after major resection surgery. This is one of the few centres in the world that have done significant numbers of function restoring surgeries, and are recognised as experts in this field, having published the protocol for functional reconstruction in the Journal of Bone and Joint Surgery and in the book Reconstructive Surgery of the Lower Extremity.

Procedures for functional restoration include Quadriceps reconstruction (to restore knee extension) - this is the most common type of functional lower limb reconstruction. Hamstring transfers were originally described for use in polio over a century ago, sartorius transfers, and free functional muscles transfers such as the latissimus dorsi or contralateral rectus femoris/ vastus lateralis.

Other techniques for functional reconstruction include anterior leg compartment reconstruction (to restore foot dorsiflexion/ prevent foot-drop) and posterior leg compartment reconstruction (to restore plantar-flexion). Techniques such as the free functional anterolateral thigh - rectus femoris muscle combined flap are also used.

Previous studies have not provided objective proof of restoration of gait, and have been limited to scores such as the Musculoskeletal Tumor Society Score (MSTS), range of motion, and Medical Research Council (MRC) grade power. These scores are of limited value in establishing whether a patient's gait is normal, and may be subject to investigator bias.

Two objective techniques will be used to assess normality of gait after functional reconstruction:

1. Three-dimensional clinical gait analysis (3DCGA) provides a robust and objective technique for measurement of how an individual walks both for clinical use and for research purposes.
2. Environmental Simulator (the Motek system at Strathclyde University): this is the only environmental simulator of its type out-with the Ministry of Defence in the United Kingdom. It provides simulated environments on a large projected screen with the patient attached to a safety harness, whilst walking on an adjustable treadmill. This allows simulation of urban environments, negotiation of trip hazards, walking up hills and shopping tasks. This will permit more tangible answers regarding the objective return to function of patients in an environmental context that they can understand eg "Will I be able to go hillwalking?" "Will I be safe to go shopping without crutches or a brace?".

Aim/Primary and Secondary Objectives

The aim of this study is to objectively assess the normality of gait after functional reconstructive surgery, and to assess whether patients can return to activities of daily living using the Environmental simulator

Methodology

Patients who have undergone functional reconstructive surgery will be identified from a prospectively held database. The patients will be invited to participate by letter and given an information sheet. Should the patient wish to participate in the study they will be invited to clinic to discuss the study with the senior researcher (SL) and sign a consent form related to gait analysis and the environmental simulator.

There are 3 components to the study:

1. Patient Reported Outcome Measurements - using validated questionnaires including the Toronto Extremity Salvage Score (TESS). Clinical assessment will include MRC grade power and range of motion.
2. 3D Gait analysis - this employs 3D cameras and pressure sensors to objectively assess the patient's ability to walk, and can identify subtle differences in gait that cannot be identified on questionnaires or on simple video analysis. Electromyography may be used to assess active muscle contraction as part of the gait analysis.
3. Environmental simulator - this will employ a state-of-the-art simulator that can assess a patient's ability to navigate simulated environments eg walking up a hill, navigating an urban environment, and shopping tasks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone major surgery for tumour, resulting in significant muscle loss in the West of Scotland
* At least 3 months post-surgery

Exclusion Criteria:

* Patients with ongoing surgical complications
* < 3 months post-surgery
* Patients currently undergoing radiotherapy
* Patients with known motion sickness (related to Virtual Reality component of gait analysis)

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Population study groups will be taken from the Scottish Sarcoma Network Glasgow centre's patient cohort
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Gait Profile Score (GPS) | Up to 10 years after surgery. From date of surgery, but after completion of post-operative rehabilitation at 6 months up to 10 years following surgery
  Objective score from 3D Gait Analysis. This is a continuous score with no minimum or maximum score, where lower scores indicate better gait.

SECONDARY OUTCOMES:
Environmental Simulator assessment of ability to complete Tasks of Daily Living | Up to 10 years after surgery. From date of surgery, but after completion of post-operative rehabilitation at 6 months up to 10 years following surgery
  Descriptive outcome measure on ability to complete simulator tasks which replicate activities of daily living.
Toronto Extremity Salvage Score (TESS) | Up to 10 years after surgery. From date of surgery, but after completion of post-operative rehabilitation at 6 months up to 10 years following surgery
  Patient reported outcome measure on function after surgery. This is a continuous score which is converted to a 0 to 100 score. Higher indicates better functional outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Canniesburn Regional Plastic Surgery and Burns Unit, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on reasonable written request